CLINICAL TRIAL: NCT07027579
Title: The Effect of Nutrition Education Program on the Quality of Life and Chronic Disease Adaptation in Patients With Thyroid Dysfunction
Brief Title: Effect of Nutrition Education on the Quality of Life, Chronic Disease Adaptation in Patients With Thyroid Dysfunction
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Çanakkale Onsekiz Mart University (Other)
Responsible Party: Principal Investigator, Naile ALANKAYA, Assoc. Prof, Çanakkale Onsekiz Mart University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: COMU-SBF-NA-03
Record Dates: First submitted 2025-06-11; First posted 2025-06-18 (Actual); Last update posted 2025-06-18 (Actual); Status verified 2025-06

CONDITIONS: Thyroid Disease
Keywords: Thyroid Dysfunction; Quality of Life; Chronic Disease Adaptation; Nutrition Education Program
MeSH Terms: conditions — Thyroid Diseases | interventions — Nutrineal; Nutrition Assessment

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervetion group (Experimental): The intervention group will consist of 30 people. Participants in the experimental group selected by appointment will receive a one-on-one face-to-face outpatient clinic training room with a power point presentation prepared by the researcher on "Nutrition for Thyroid Patients" and a computer. At the end of the training, a "Nutrition for Thyroid Patients" training booklet will also be given.The education will be delivered as a single session, with an expected duration of approximately 30-35 minutes. Following the training, the Nutrition Attitude Scale, Chronic Illness Adherence Scale (CIAS) and Quality of Life Scale for Thyroid Patients (ThyPRO) will be re-administered to reassess participants' knowledge levels.
  Interventions: Other: Nutrineal
- Control group (No Intervention): The control group will consist of 30 people. All patients will be asked to complete the Nutrition Attitude Scale, Quality of Life Scale for Thyroid Patients (ThyPRO) and Chronic Illness Adherence Scale (CIAS). Patients in the control group will not receive any training. The same forms will be filled out for the final test 3 months later. Patients who wish to will be given the training provided in the experimental group.

INTERVENTIONS:
Other: Nutrineal — The "Education for Thyroid Patients' Nutrition" power point presentation prepared by the researcher will also be done using a computer.
  Other Names: Nutrition Education
  Arms: Intervetion group

SUMMARY:
This thesis study is designed to examine the effects of nutrition education provided to individuals with thyroid dysfunction on their quality of life and adaptation to the disease. The data will be collected using the Descriptive Characteristics Form, the Nutrition Attitude Scale, the Quality of Life Scale for Thyroid Patients (ThyPRO), and the Chronic Illness Adherence Scale. The Body Mass Index (BMI) of participating patients will be calculated by the researcher based on measured height and weight. Laboratory values including TSH, free T4, and free T3 will be obtained from the patients' medical records on the day of assessment. Data collection will be conducted in two phases. The study population will consist of all patients diagnosed with thyroid dysfunction who present to Dr. Burhan Nalbantoğlu Hospital. Using the G*Power 3.1.9.2 software, the required sample size was calculated prior to data collection with a 95% confidence level. For correlation analysis, an alpha value of 0.05, an effect size of 0.455, and a statistical power of 95% were assumed, resulting in a minimum sample size of 56 participants (30 per group). Accounting for potential data loss, a total of 60 patients (30 per group) are planned to be included in the sample.

DETAILED DESCRIPTION:
This thesis study is designed to examine the effects of nutrition education provided to individuals with thyroid dysfunction on their quality of life and adaptation to the disease. Patients with thyroid disorders are affected both physically and socially due to hormonal imbalances. In this context, the study aims to investigate how dietary habits are shaped and how these habits influence individuals' overall quality of life. Accordingly, the following research questions were addressed:

* Does the nutrition education provided affect the level of nutritional knowledge in patients with thyroid dysfunction?
* Does the nutrition education provided improve the quality of life in patients with thyroid dysfunction?
* Does the nutrition education provided enhance disease adaptation in patients with thyroid dysfunction? Implementation of the Study Prior to the nutrition education, patients will be informed about the purpose of the study, the data collection methods, and the content of the educational topics. Patients who agree to participate in the study will be asked to sign an informed consent form. The Body Mass Index (BMI) of participating patients will be calculated by the researcher based on measured height and weight. Laboratory values including TSH, free T4, and free T3 will be obtained from the patients' medical records on the day of assessment. Data collection will be conducted in two phases.

Phase 1:

All patients who agree to participate in the study (both intervention and control groups) will first be asked to complete the "Descriptive Characteristics Form," the "Nutrition Attitude Scale" to assess their dietary habits, the "ThyPRO Questionnaire" to evaluate thyroid-related quality of life, and the "Chronic Illness Adherence Scale (CIAS)" to assess disease adaptation.

The Body Mass Index (BMI) of each participant will be calculated by the researcher through direct measurement of height and weight. Free T4 and free T3 values will be obtained from the patients' medical records on the day of evaluation.

Participants in the intervention group, selected through randomization, will receive a one-on-one, face-to-face educational session in the outpatient clinic's education room. The session will be conducted by the researcher using a PowerPoint presentation titled "Nutrition Education for Thyroid Patients," prepared specifically for the study and delivered via computer. At the end of the session, participants will also be provided with a printed "Nutrition Guide for Thyroid Patients." Participants in the control group will not receive the educational session at this stage; however, they will be given the same printed "Nutrition Guide for Thyroid Patients" prepared by the researcher. It will be communicated to the control group that the same individual training session will be offered to them after the study concludes.

The education will be delivered as a single session, with an expected duration of approximately 30-35 minutes. Following the training, the "Nutrition Attitude Scale" will be re-administered to reassess participants' knowledge levels.

Phase 2:

Three months after the initial planned education session, participants will again complete the "Nutrition Attitude Scale" to assess changes in dietary habits, as well as the "ThyPRO Questionnaire" and the "Chronic Illness Adherence Scale (CIAS)" to evaluate changes in thyroid-related quality of life and disease adaptation. If available, free T4 and free T3 values will be obtained from hospital records on the day of follow-up, and BMI will be recalculated by the researcher.

Participants in the control group will also be asked to complete the same forms three months after the initial assessment. Following the completion of the data collection process, the same one-on-one education provided to the intervention group will be delivered to the control group to eliminate any disadvantage or ethical concerns.

Data Collection Tools:

The data will be collected using the Descriptive Characteristics Form, the Nutrition Attitude Scale, the Quality of Life Scale for Thyroid Patients (ThyPRO), and the Chronic Illness Adherence Scale.

The study population will consist of all patients diagnosed with thyroid dysfunction who present to Dr. Burhan Nalbantoğlu Hospital. Using the G*Power 3.1.9.2 software, the required sample size was calculated prior to data collection with a 95% confidence level. For correlation analysis, an alpha value of 0.05, an effect size of 0.455, and a statistical power of 95% were assumed, resulting in a minimum sample size of 56 participants (30 per group). Accounting for potential data loss, a total of 60 patients (30 per group) are planned to be included in the sample.

Data Analysis The data obtained in the study will be analyzed using SPSS software (Windows version 25.0). Descriptive statistical methods such as frequency, percentage, minimum-maximum values, median, mean, and standard deviation will be used for data evaluation. The normality of the data for the scales used will be assessed through tests of skewness and kurtosis. For normally distributed quantitative data, comparisons between two independent groups will be performed using the independent samples t-test, while comparisons among more than two groups will be conducted using one-way analysis of variance (ANOVA).

ELIGIBILITY:
Inclusion Criteria:

* Not having any physical or mental disabilities
* Not having received such training before
* Volunteering to participate in the study
* Be 18 years of age or older.

Exclusion Criteria:

* Being under 18 years of age.
* Having cognitive dysfunction.
* Not volunteering to participate in the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2025-07-20 (Estimated); Primary Completion 2025-09-15 (Estimated); Study Completion 2025-12-30 (Estimated)

PRIMARY OUTCOMES:
Quality of Life Scale for Thyroid Patients (ThyPRO) | Baseline and after 6 months
  The "Thyroid-Related Quality of Life Questionnaire - ThyPRO" consists of 12 items. The 12th question stands alone and is analyzed separately. The scale does not yield a total score; instead, each subscale is scored individually on a scale ranging from 0 to 100. Higher scores indicate lower quality of life.
Nutrition Attitude Scale | Baseline and after 6 months
  The Nutrition Attitude Scale (NAS) is a five-point Likert-type scale rated from "Strongly agree" (5) to "Strongly disagree" (1). The scale consists of 21 items in total-20 positive and 1 negative. The lowest 21 points and the highest 105 points can be obtained from the nutrition attitude scale. Higher scores from the scale; It will reveal that the individuals who filled the scale have a high attitude towards nutrition and those who have low scores have a low attitude towards nutrition. It can be asserted that individuals' high attitude scores towards nutrition are sensitive to weight control and health.
Chronic Illness Adaptation Scale (CIAS) | Baseline and after 6 months
  The scale consists of 25 items across three sub-dimensions: physical adaptation, social adaptation, and psychological adaptation.The total possible score on the scale is 125. Higher scores on the sub-dimensions and/or the total scale indicate a greater level of adaptation to the disease.

CONTACTS AND LOCATIONS:
Overall Officials: NAİLE ALANKAYA, Assoc. Prof, Study Director — Çanakkale Onsekiz Mart University, Faculty of Health Sciences
Locations (1):
- Çanakkale Onsekiz Mart University, Faculty of Health Sciences, Çanakkale, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No